CLINICAL TRIAL: NCT01465594
Title: Randomized Study Comparing Urinary Diversion by Suprapubic Catheter With Transurethral Catheter in Patients After Radical Prostatectomy
Brief Title: Study Comparing Urinary Diversion (Transurethral/Suprapubic) After Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: catheterstudy001
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Pain; Catheter Complications
Keywords: Pain Measurement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- transurethral catheter after EERPE/ RALP (Active Comparator): Recording of QoL measured by visual analogue ( pain )scale,EORTC QlQ -C 30 and QLQ - PR 25 questionnaires, incontinence rate, complication rate regarding insufficiency and strictures of vesicourethral anastomoses and urinary tract infection; demand of re-catheterization due to urinary retention and demand of antispasmodics
  Interventions: Procedure: transurethral catheter after EERPE/ RALP; Procedure: suprapubic catheter after EERPE /RALP
- suprapubic catheter after EERPE /RALP (Active Comparator): Recording of QoL measured by visual analogue ( pain )scale,EORTC QlQ -C 30 and QLQ - PR 25 questionnaires, incontinence rate, complication rate regarding insufficiency and strictures of vesicourethral anastomoses and urinary tract infection; demand of re-catheterization due to urinary retention and demand of antispasmodics
  Interventions: Procedure: transurethral catheter after EERPE/ RALP; Procedure: suprapubic catheter after EERPE /RALP

INTERVENTIONS:
Procedure: transurethral catheter after EERPE/ RALP — transurethral catheter after EERPE/ RALP
Procedure: suprapubic catheter after EERPE /RALP — suprapubic catheter after EERPE /RALP

SUMMARY:
The study aims to show the technical feasibility of the suprapubic urinary diversion after endoscopic extraperitoneal radical prostatectomy (EERPE) and has a greater comfort for the patients with at least the same catheter complication rate in comparison to the urethral urinary diversion.

DETAILED DESCRIPTION:
Patients are randomized 1:1 in the different arms Recording of QoL measured by visual analogue ( pain )scale,EORTC QlQ -C 30 and QLQ - PR 25 questionnaires, incontinence rate, complication rate regarding insufficiency and strictures of vesicourethral anastomoses and urinary tract infection; demand of re-catheterization due to urinary retention and demand of antispasmodics

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate,
* Subjects treated by conventional or robotic assisted laparoscopic prostatectomy
* Be willing/able to adhere to follow up visits

Exclusion Criteria:

* Subjects treated by retropubic or perineal prostatectomy Subjects with known bladder cancer
* Contraindications for anticholinergic drugs
* Waist measurement > 100 cm
* No written informed consent
* Age < 18 years
* Subjects with known narrow-angle glaucoma

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Superiority of suprapubic catheter after EERPE | 2nd postoperative day
  Superiority of suprapubic catheter versus transurethral catheter regarding QoL /Patient comfort

SECONDARY OUTCOMES:
Comparison of QoL in both arms measured by visual analogue (pain) scale | 1st and 3rd until 5th postoperative day
  Comparison of QoL in both arms measured by visual analogue (pain) scale, EORTC QlQ -C 30 and QLQ - PR 25 questionnaires, incontinence rate, complication rate regarding insufficiency and strictures of vesicourethral anastomoses and urinary tract infection; demand of re-catheterization due to urinary retention and demand of antispasmodics.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Arsov, Dr, Principal Investigator — Heinrich Heine Universität
Locations (1):
- University Hospital, Urological department, Düsseldorf, Germany